CLINICAL TRIAL: NCT03747718
Title: A Study for Evaluation of Clinical Response to Single vs. Maintenance Fecal Microbiota Transplantation in Pediatric Patients With Refractory Crohn's Disease
Brief Title: Randomized Trial Comparing Single vs. Maintenance Fecal Microbiota Transplant for Refractory Crohn's Disease in Children
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Alka Goyal, Clinical Professor of Pediatrics, Stanford University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: CMH-17010048
Record Dates: First submitted 2018-03-08; First posted 2018-11-20 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Crohn Disease
Keywords: Crohn's; Pediatric; IBD; Fecal
MeSH Terms: conditions — Crohn Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: The study will operate as a single group open label study until visit 6, at which point it will become a randomized trial.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking will be completed at the 1.5 month visit by the pharmacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fecal Microbiota Follow up Enemas (Experimental): In this arm subjects will receive 3 fecal microbiota transplants at 1 monthly intervals at 1.5, 2.5 and 3.5 months (+/- 2 weeks) after transplant
  Interventions: Biological: Fecal Microbiota Transplantation
- Placebo Enemas (Placebo Comparator): In this arm subjects will receive 3 placebo transplants at 1 monthly intervals at 1.5, 2.5 and 3.5 months (+/- 2 weeks) after transplant
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Fecal Microbiota Transplantation — Fecal Microbiota Transplantation via colonoscopy for the first transplant in all subjects. This will be followed by 2 fecal enema transplants for all subjects 7 days (+/- 3 days) after colonoscopy. All subjects will be assessed 1.5 months (+/- 2 weeks) after colonoscopy. The subjects who are deemed responders based on a drop in PCDAI=12.5 or higher will be randomized to receive fecal or placebo enemas at 1 monthly (+/- 2 weeks) enemas at 1.5, 2.5 and 3.5 months after colonoscopy. All subjects will be assessed at 4.5 and 6 months (+/- 2 weeks) following colonoscopy. The study will be completed at 6 months (+/- 2 weeks) following colonoscopy.
  Arms: Fecal Microbiota Follow up Enemas
Other: Placebo — Fecal Microbiota Transplantation via colonoscopy for the first transplant in all subjects. This will be followed by 2 fecal enema transplants for all subjects 7 days (+/- 3 days) after colonoscopy. All subjects will be assessed 1.5 months (+/- 2 weeks) after colonoscopy. The subjects who are deemed responders based on a drop in PCDAI=12.5 or higher will be randomized to receive fecal or placebo enemas at 1 monthly (+/- 2 weeks) enemas at 1.5, 2.5 and 3.5 months after colonoscopy. All subjects will be assessed at 4.5 and 6 months (+/- 2 weeks) following colonoscopy. The study will be completed at 6 months (+/- 2 weeks) following colonoscopy.
  Arms: Placebo Enemas

SUMMARY:
NCT02108821

Primary goal:

-To determine the safety of fecal transplant by colonoscopy and retention enemas for induction followed by maintenance retention fecal vs. placebo enemas in children and young adults with uncomplicated mild-moderately active Crohn's disease.

Secondary goals:

* Assess efficacy of this induction regimen followed by maintenance fecal or placebo transplants in responders. The efficacy will be assessed by clinical evaluation and fecal calprotectin that is a non-invasive biomarker.
* Correlate subject's baseline microbiome findings with likelihood for response to FMT induction therapy.
* Follow the chronological microbiome shifts after transplant and correlate with response using clinical and calprotectin assessment in the two groups.

DETAILED DESCRIPTION:
NCT02108821 Detailed Description: Gut microbiome plays a key role in gut immunology and function. A disturbance in the diversity of gut bacterial composition could be linked to several immune mediated diseases including Inflammatory Bowel Diseases IBD. IBD can be classified into Crohn's Disease CD, Ulcerative Colitis UC and indeterminate colitis IC, these diseases occur from an aberrant immune reaction to resident gut bacteria. CD can affect the entire gut in a transmural fashion whereas UC involves primarily the mucosal layer of the colon. The treatment options often overlap in both conditions. It has also been demonstrated that both recurrent Clostridium difficile infection RCDI and IBD are associated with gut dysbiosis. The process of fecal microbiota transplantation FMT, where fecal microbial community from a healthy individual is transferred into a recipient, has been established as an efficacious therapy for RCDI.

The role of FMT in treatment of IBD is still not well established. Recent data on FMT in UC has shown promising results. Three out of the four double blind randomized trials demonstrated superiority of FMT compared to placebo. The first randomized trial was conducted by Moayyedi et al. in which six weekly fecal or water placebo enemas demonstrated a remission rate in 24 percent vs. 5 percent in fecal and placebo group respectively which was found to be statistically significant 1. Similarly FMT was found to be superior to placebo in achieving clinical remission at week 8 2 percent FMT vs. 8 percent placebo by Paramsothy et. al who gave fecal or placebo enemas 5 days a week for 8 weeks 2. Costello et. al used multidonor fecal suspension compared to placebo autologous stool via colonoscopy followed by 2 retention enemas by day 7. They observed a significantly superior rate of remission 32 percent vs. 9 percent with fecal and placebo enemas respectively 3. Rossen et. al reported results of FMT in UC where they used two nasoduodenal infusions, 3 weeks apart with no significant benefit in the group that received fecal infusions compared to the placebo 4. There have been no published randomized trials for CD. An open label study on pediatric CD by Suskind et al showed promising results with response in 7 out of 9 children with a single fecal transplant delivered by nasogastric tube 5. Another open-label study of 30 CD adult patients who received a single FMT into the small bowel demonstrated 86.7 percent clinical improvement in the first month after transplant that was sustained in 66.7 percent patients till 6 months 6. A recent meta-analysis on FMT as a primary or adjunct therapy for IBD in cohort studies showed clinical remission in 22 percent and 60.5 percent patients with UC and CD respectively. It was found to be a safe procedure in both conditions. The authors also speculated that children with IBD might respond better to FMT compared to adult patients 7.

Data on FMT in UC has thus demonstrated better results when multiple enemas are used for induction. So far results from open-label studies on Crohn's disease also look promising. However there is still a gap in knowledge and understanding about the safety, outcome and preferred route of FMT for induction of remission in Crohn's disease. Additionally, the role or frequency of maintenance therapy with retention enemas has not been studied.

In this proposed randomized trial, the investigators will perform an open-label induction with fecal transplantation on the subjects with medically refractory mild to moderately active but Clostridium Difficile CDI negative and otherwise uncomplicated Crohn's disease. Subjects who meet the inclusion criteria will receive the initial FMT into right colon while undergoing a medically indicated colonoscopy. This will be followed by 2 retention enemas at 1 and 2 weeks plus 3 days after colonoscopy as long as they are able to tolerate this treatment. All subjects will then be assessed at 6 weeks for response to FMT that will be defined by a drop in PCDAI by 12.5 points. The responders will be randomized to fecal vs. placebo maintenance retention enemas at 1-monthly intervals for 3 months. The subjects will be followed for 6 months from the initial colonoscopy to assess for medium-term outcome and response.

Primary goal:

-To determine the safety of fecal transplant by colonoscopy and retention enemas for induction followed by maintenance retention fecal vs. placebo enemas in children and young adults with uncomplicated mild-moderately active Crohn's disease.

Secondary goals:

* Assess efficacy of this induction regimen followed by maintenance fecal or placebo transplants in responders. The efficacy will be assessed by clinical evaluation and fecal calprotectin that is a non-invasive biomarker.
* Correlate subject's baseline microbiome findings with likelihood for response to FMT induction therapy.
* Follow the chronological microbiome shifts after transplant and correlate with response using clinical and calprotectin assessment in the two groups.

All subjects will maintain an adverse event diary and will be assessed 1 week after each transplant either on telephone or in the clinic. They will have access to the medical providers for 24 hours a day including weekends. They will also be assessed in the clinic prior to each transplant procedure and at 6 months following colonoscopy. Blood work for blood counts CBC with Diff, erythrocyte sedimentation rate ESR, C reactive protein CRP, liver function tests LFTs If clinically Indicated and fecal calprotectin will be assessed at baseline, as well as at 1.5 and 6 months (+/- 2 weeks) after initial colonoscopy for FMT. Stool collection for microbiome analysis will be performed at baseline and subsequently at 1.5, 3.5 and 6 months (+/- 2 weeks) following initial colonoscopy.

Thirty subjects who are 2-25 years of age at the time of consenting will be enrolled in the trial over a period of 24 months. Subjects with mild-moderate Crohn's disease defined as having Pediatric Crohn's Disease Activity Index PCDAI of 10-37.5 despite standard medical therapy that has been stable for at least 4 weeks and are undergoing a medically indicated colonoscopy will be eligible for screening. All enrolled subjects will get FMT via colonoscopy into the right colon along with routine biopsies. Additional biopsies will be collected from the terminal ileum and rectum for microbiome analysis and also stored for future studies. Microbiota analysis will be performed on the donor at the time of stool collection by Open-Biome and recipient stool sample collected within 7 (+/- 3 days) days prior the scheduled fecal microbiota transplantation. They will be followed for adverse events throughout the duration of the study. The clinical response will be defined as a drop in PCDAI by 12.5 points. The clinical response and fecal microbiome changes will be assessed at 1.5, 2.5, 3.5 and 6 month (+/- 2 weeks) throughout the duration of the study. The subjects assessed as responders at 1.5-month will be randomized to receive monthly maintenance retention fecal or placebo enemas for 3 consecutive months. The enrolled subjects will have blood work CBC with diff, ESR, CRP, LFTs and fecal calprotectin evaluation at baseline, 1.5 and 6 months (+/- 2 weeks). The investigators will utilize the Open-Biome laboratory as the fecal stool bank to supply both placebo and fecal suspension for transplant. The investigators estimate that they will screen up to 100 patients with Crohn's Disease CD over 2 years, to reach our goal of 30 total study participants. Subjects who do not improve at 1.5 month post transplant assessment or require prompt intervention at any time during this study will be offered escalation of medical therapy. All subjects will be clinically assessed at 1.5, 2.5, 3.5, 4.5 and 6 months (+/- 2 weeks) post colonoscopy. A rescue retention enema will be allowed during the study if a subject who was previously responding develops a flare.

The investigators hypothesize that fecal transplant will be a safe therapy in uncomplicated mild-moderate Crohn's disease patients. About 60 percent of the subjects are likely to respond at 1.5 month assessment. Subjects receiving maintenance fecal transplants will have a longer duration of remission compared to those who receive only the induction treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects between the age of 2 and 25 years.
2. Current CD patients who have either:

   o CD with mild to moderately active disease (PCDAI 10-37.5) due to failure of current therapy that has been stable for 4 weeks and are undergoing colonoscopy. For this study we will recruit only those CD patients who have disease only in colon or colon and terminal ileum so disease can be accurately assessed prior to and after FMT.
3. The ability to safely undergo colonoscopy (physical status classification of one through three used by the American Society of Anesthesiologists, see Appendix A) as determined by Principal Investigator.
4. Females of childbearing potential must have a negative urine pregnancy test during screening and a negative urine pregnancy test at visit 2 (FMT procedure day).
5. Informed consent and assent (per IRB/EC), as appropriate.
6. Subject must be willing to comply with all study related procedures, follow up visits and complete home diaries.

Exclusion Criteria:

1. Severe immunosuppression: concomitant steroids (1mg/kg/day or greater than 30 mg/day) and biologicals like infliximab, Adalimumab, Golimumab, Certolizuman, Ustekinemab.
2. Neutropenia (500 neutrophils/mL) or other severe immunosuppression. Anti-TNF will be permitted. Patients on monoclonal antibodies to B and T cells, calcineurin inhibitors (tacrolimus, cyclosporine) and mycophenolate mofetil may be enrolled only after consultation with the medical monitor.
3. Established central line or planned placement during trial.
4. Pressor or ventilator support.
5. On antibiotics with the inability to discontinue within 4 weeks prior to FMT procedure.
6. Requires continued antibiotic use or anticipates antibiotic use in upcoming 4 weeks.
7. Patients found to have complications such as an abscess, phlegmon, stricture, small bowel obstruction, perforation, internal or external fistulation or infection as causes for flare up.
8. Not willing or able to consent or follow guidelines throughout research trial.
9. Non-English Speaking
10. Worsening Inflammatory Bowel disease between time of consenting and FMT resulting in PCDAI greater than 40, or are unable to wait for the routine procedure due to rapid deterioration.
11. A condition that would jeopardize the safety or rights of the subject, would make it unlikely for the subject to complete the study, or would confound the results of the study
12. Participation in an investigational drug study within 30 days of screening.
13. Change in therapy within the previous 30 days.
14. Female patients of childbearing age who are pregnant, lactating, or plan to become pregnant during study.
15. Active or gastrointestinal infection at time of enrollment.
16. Known or suspected toxic megacolon
17. Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment. This does not include appendectomy or cholecystectomy.
18. Admitted to or expected to an intensive care unit for medical reasons (not just boarding).
19. Concurrent intensive induction chemotherapy, radiation therapy or biological treatment for active malignancy. Patients on maintenance chemotherapy may be enrolled only after consultation with medical monitor
20. Expected life expectancy less than 6 months
21. Previous usage of FMT products within 1 year of enrollment excluding this study.
22. Patients with a history of severe anaphylactic or anaphylactoid food allergy.
23. Solid organ transplant recipients 90 days post-transplant or on active treatment for rejection.
24. If at risk for CMV associated disease (at investigator's discretion, e.g. immunocompromised), negative IgG testing for cytomegalovirus (CMV).
25. Severe anal fissues.
26. Stool infections including C.Diff (checked at the study center for consistency). If positive for C.Diff, they can be eligible if symptoms persist despite successful treatment and negative stool test obtained 1 month after discontinuation of antibiotics.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by Adverse events | 6 months
  The symptom diary will be used for the subject to document any adverse events that occur during the trial. This will be reviewed at each study visit. Number of participants with treatment related adverse events as assessed by CTCAE v 4.0

SECONDARY OUTCOMES:
Efficacy as assessed by Physician Global Assessment (PGA) | 6 months
  The PGA will be recorded during the study at baseline, 1.5, 2.5, 3.5, 4.5 and 6 months (+/- 2 weeks) to measure efficacy of treatment over time.
Efficacy as assessed by PCDAI (Pediatric crohn's disease Activity Index)analysis | 6 months
  The PCDAI will be completed at each study visit at baseline, 1.5, 2.5, 3.5, 4.5 and 6 months (+/- 2 weeks) to assess efficacy of treatment.
Response as assessed by fecal calprotectin | Calprotectin will be measures at baseline, 1.5 month and 6 months (+/- 2 weeks) after transplantation
  Fecal calprotectin is a non invasive marker for colon inflammation
Response as assessed by fecal microbiota changes | Microbiome will be measures at baseline, 1.5, 3.5 and 6 months (+/- 2 weeks) after transplantation
  Diversity and structure of Fecal microbial community will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Alka Goyal, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States